CLINICAL TRIAL: NCT01998646
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Dose Escalation Study to Assess the Safety, Tolerability, and Pharmacoknetics of ASP4058 Following Single Oral Doses in Healthy Subjects
Brief Title: A Dose Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of ASP4058 Following Single Oral Doses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 4058-CL-1001
Record Dates: First submitted 2013-11-25; First posted 2013-12-02 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-11

CONDITIONS: Pharmacokinetics of ASP4058; Healthy Subjects; Food Effect of ASP4058
Keywords: ASP4058; healthy subjects
MeSH Terms: interventions — ASP4058

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ASP4058 Tablet Dose Escalation Cohort (Experimental)
  Interventions: Drug: ASP4058
- ASP4058 Tablet - Fasting conditions (Experimental)
  Interventions: Drug: ASP4058
- ASP4058 Tablet - Fed conditions (Experimental)
  Interventions: Drug: ASP4058
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP4058 — Oral tablet
  Arms: ASP4058 Tablet - Fasting conditions; ASP4058 Tablet - Fed conditions; ASP4058 Tablet Dose Escalation Cohort
Drug: Placebo — Oral tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to explore the safety, tolerability and pharmacokinetics (PK) of single ascending oral doses of ASP4058 in non-elderly, healthy male and female subjects. This study will also explore the effect of food on the PK of ASP4058.The food-effect crossover group was open-label treatment with no placebo control.

DETAILED DESCRIPTION:
Subjects will remain in the clinic for 9 days. Subjects will return to the clinic for follow-up on days 12 and 30 to collect additional safety information.

ELIGIBILITY:
Inclusion Criteria:

* The female subject must be at least two years postmenopausal (defined as at least 2 years at Screening without menses and a confirmatory follicle stimulating hormone (FSH) level of ≥ 40 U/L at Screening) or surgically sterile (with documentation provided by a healthcare professional) and not pregnant or lactating.
* The male subject agrees to sexual abstinence, is surgically sterile (with documentation provided by a healthcare professional), or is using a medically acceptable method (e.g., spermicide and diaphragm, or spermicide and condom) to prevent pregnancy and agrees to continue using this method until end of study or 29 days post-dose, whichever is longer.
* The subject must have normal (≥ 80% of normal range) respiratory function as defined by spirometry, measuring forced expiratory volume (FEV1) and forced vital capacity (FVC) relative to established normal ranges adjusted for age and sex.
* The subject at Screening and Day -2, must have color vision testing, acuity testing (corrected), and a fundoscopic exam that are within normal limits in the opinion of the examining/reviewing ophthalmologist.
* The subject's total lymphocyte count at Screening must be >1.0 x 103/uL.
* The subject is highly likely to comply with the protocol-defined procedures and complete the study.
* The subject is positive for herpes simplex virus (HSV)-1 and/or HSV-2 anti-bodies at Screening.

Exclusion Criteria:

* The subject is a current smoker or has a history of routinely smoking (>10 cigarettes/day) within the last seven years..
* The subject has a history of clinically significant bradyarrhythmia or sinus bradycardia.
* The subject has any condition possibly affecting drug absorption (e.g., gastrectomy).
* The subject has history of consuming more than 14 units of alcoholic beverages per week on average within 6 months prior to Screening or has a history of alcoholism or drug/chemical/substance abuse within past 2 years prior to Screening or the subject tests positive at Screening or clinic admission for alcohol or drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, and opiates).
* The subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 2 weeks prior to clinic check in.
* The subject has a supine mean systolic blood pressure < 90 or > 140 mmHg and a mean diastolic blood pressure < 50 or > 90 mmHg, or mean heart rate > 100 or < 55 beats per minute (bpm), either at Screening or clinic check in (measurements taken in triplicate after subject has been resting in a supine position for a minimum of 5 minutes).
* The subject has 12-lead electrocardiogram (ECG) demonstrating QTcF > 450 msec (female) or > 430 msec (male) at Screening. If QTcF exceeds the limits above, the ECG should be repeated two more times and the average of the three QTcF values should be used to determine the subject's eligibility.
* The subject has been diagnosed with glaucoma or is currently being treated for glaucoma.
* The subject is known to be positive for human immunodeficiency virus (HIV) antibody.
* The subject is currently using Latisse® (eyelash lengthening medication) or has used it within the last 30 days.
* The subject has a positive test for hepatitis C antibody (HCV), or positive for hepatitis B antigen (HBsAg) at Screening.
* The subject has used prescription or non-prescription drugs within 2 weeks or 5 half lives (whichever is longer) or complementary and alternative medicines (CAM) within 28 days prior to study drug administration (excluding hormone replacement therapy [HRT] and acetaminophen).
* The subject has participated in a clinical trial and received an experimental agent or has participated in a clinical trial of approved therapy for investigational use within 30 days or ten half-lives, whichever is longer, prior to study drug administration.
* The subject has been vaccinated within the last 60 days.
* The subject has had any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or has donated plasma within 7 days prior to clinic admission on Day -2.
* The subject is known positive for tuberculosis or has tested positive at Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2010-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter of ASP4058: Cmax | Day 1-8
  Maximum Concentration (Cmax)
Pharmacokinetic parameter of ASP4058: AUCinf | Day 1-8
  Area Under the Concentration - Time curve from time 0 extrapolated to infinity (AUCinf)

SECONDARY OUTCOMES:
Composite of pharmacokinetic parameters of ASP4058 in plasma: AUClast, Tmax, t1/2, tlag, Vz/F, CL/F | Day 1-8
  Area Under the Concentration - Time curve from time 0 up to the last quantifiable concentration (AUClast), Time to Attain Cmax (Tmax), Apparent Terminal Elimination Half-life (t1/2), Time prior to the first measurable (non-zero) concentration (tlag), Apparent Volume of Distribution During the Terminal Phase of the Plasma Concentration vs. Time Profile (Vz/F), Apparent Total Body Plasma Clearance (CL/F)
Composite of pharmacokinetic parameter of ASP4058 in urine: Aelast, Aelast%, CLr | Day 1-8
  Cumulative urine drug excretion from time 0 up to the last measurable concentration (Aelast), Fraction of drug into urine up to the collection time of the last measurable concentration (Aelast%), Renal Clearance (CLr)
Pharmacodynamics of ASP4058: white blood cell determination with differentials, lymphocyte subsets | Day 1-8

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami, Inc, Miami, Florida
  - Covance Clinical Research Unit, Inc., Evansville, Indiana